CLINICAL TRIAL: NCT03905356
Title: Exercise Therapy in Radiation Therapy (EXERT)
Brief Title: Exercise Therapy in Radiation Therapy
Acronym: EXERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Kathleen Sturgeon, Assistant Professor, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00010618
Record Dates: First submitted 2019-03-28; First posted 2019-04-05 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): The exercise intervention will utilize the "Moving Through Cancer: A Guide to Exercise for Cancer Survivors" framework. A certified cancer exercise physiologist will work through this guide at radiation therapy visits, with at least 1 visit per week, per the study schema. The cancer exercise physiologist will teach participants proper: warm ups, use of equipment, exercise form, modes of activity, intensity of exercise, flexibility exercises, and cool down. The cancer exercise physiologist will tailor the instruction to convey special considerations for exercise based on treatment and cancer type. The patient will perform supervised exercise in the Exercise Medicine Unit under the guidance of the cancer exercise specialist. The exercise done will be educational in nature (i.e. learning about proper walking form, proper intensity for a warmup/cool down, proper techniques for resistance exercises).
  Interventions: Behavioral: Exercise Therapy

INTERVENTIONS:
Behavioral: Exercise Therapy — Certified exercise oncology specialists will personalize, prescribe, and guide ET, including twice weekly resistance training and walking, performed at home, with supervision in the Exercise Medicine Unit. The cancer exercise physiologist will teach participants proper warm ups, use of equipment, exercise form, modes of activity, intensity of exercise, flexibility exercises, and cool down. In addition, patients will be instructed to exercise on their own, at home, according to the instructions from the cancer exercise specialist.

SUMMARY:
The purpose of this study is to evaluate exercise therapy as a method for potentially improving radiation therapy treatment toxicities for metastatic cancer patients receiving radiation therapy.

DETAILED DESCRIPTION:
Study Objectives and Endpoints:

Aim 1. To determine the acceptability, feasibility, and safety of an exercise intervention among cancer patients receiving radiation therapy. The investigators anticipate that >25% of approached patients will consent to the protocol; >33% of eligible radiation therapy patients who consent will perform the exercise prescribed (based on the response rate from EnACT); and <25% of participants will experience a musculoskeletal impairment (without treatment alterations) and <5% will experience a musculoskeletal injury with symptoms lasting ≥ week or requiring medical attention. The investigators' approach will be to include patients receiving definitive RT; excluding patients at high risk for side effects from combination therapy, including fracture or cardiovascular events.

Aim 2. To discern the clinical outcomes of patients receiving RT+ET. The hypothesis is that adding ET to RT will improve patient reported outcomes and physical functioning. The investigators' approach will be to use standardized questionnaires and assessment tools: patient reported outcomes will be assessed using Common Terminology Criteria for Adverse Events - Patient Reported Outcomes (CTCAE-PROs), loaded onto tablets that patients use in the clinic. Questions will assess global PROs relevant to the ability to tolerate RT, including fatigue, pain, nausea, vomiting; and disease-site-specific PROs, including genitourinary/sexual symptoms for patients receiving pelvic RT. RT dose alterations will be documented. Scores will be compared pre- vs post- RT. The investigators will also use standardized measures already used in EnACT, including grip strength, 30-second chair stand, timed up-and-go, and 4-stage balance. Scores will be compared pre- vs post- RT.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥18 years of age
* Fluent in written and spoken English
* Must be able to provide and understand informed consent
* Must have an ECOG PS of ≤ 2
* Diagnosed with metastatic disease
* Cancer patients (stage 1-4)
* Treatment to primary site or metastatic disease
* Scheduled to receive radiation therapy at Penn State Cancer Institute
* Absence of absolute contraindications for exercise according to the American Heart Association (see below)
* Primary attending oncologist approval
* Receiving treatment as an outpatient

Exclusion Criteria:

* Receiving radiation therapy at a location other than Penn State Cancer Institute
* Not fluent in written and spoken English
* Evidence in the medical record of an absolute contraindication for exercise
* Performing > 90 minutes/week of physical activity at the time of initial evaluation
* Cardiac exclusion criteria:

  * Class II, III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty or stenting within the past 6 months prior to the start of radiation therapy
  * Uncontrolled arrhythmias; patients with rate controlled atrial fibrillation for >1 month prior to start of radiation therapy may be eligible
  * syncope
  * acute myocarditis, pericarditis, or endocarditis
  * acute pulmonary embolus or pulmonary infarction
  * thrombosis of lower extremities
  * suspected dissecting aneurysm
  * pulmonary edema
  * respiratory failure
  * acute non-cardiopulmonary disorder that may affect exercise performance or be aggravated by exercise
  * mental impairment leading to inability to cooperate
* Pregnant women
* In-patient receiving radiation therapy for a radiation emergency (e.g. cord compression, SVC syndrome, brain metastases)
* High risk of fracture or spine instability (Mirels score ≥7, SINS ≥7)
* Children (the protocol will only include individuals 18 and older)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Acceptability of exercise intervention: (number of patients agreeing to perform RT+ET)/(number approached) | 1 year
  (number of patients agreeing to perform RT+ET)/(number approached)
Feasibility of exercise intervention: (number of patients who completed RT+ET)/(number agreeing to perform RT+ET) | 1 year
  (number of patients who completed RT+ET)/(number agreeing to perform RT+ET)
Incidence of Treatment- Emergent Adverse Events | 1 year
  Safety of exercise intervention: freedom from any Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or higher event

SECONDARY OUTCOMES:
Change in timed up and go | 3 Months
  Timed up and go
change in grip strength | 3 Months
  Grip strength
change in quality of life measured via the Godin Physical Activity Questionnaire | 3 Months
  The Godin Physical Activity Questionnaire asks how much physical activity the participant engages in during a typical 7-day period.
change in quality of life measured via the Barriers to Exercise RM 5-FM survey | 3 Months
  The Barriers to Exercise RM 5-FM survey asks participants about barriers to being active. Response options include: very likely; somewhat likely; somewhat unlikely; very unlikely.
change in quality of life measured via the Work Productivity and Activity Impairment Questionnaire | 3 Months
  The Work Productivity and Activity Impairment Questionnaire ask about the effect of the participant's health problems on the ability to work and perform regular activities. A variety of question/response styles are included in the survey.
change in quality of life measured via the Scored Patient-Generated Subjective Global Assessment | 3 Months
  The Score Patient-Generated Subjective Global Assessment asks about participant nutrition. A variety of question/response styles are included in the survey.
change in quality of life measured via the EORTC questionnaire | 3 Months
  The EORTC Quality of life questionnaire asks a variety of questions about their health regarding physical abilities. Response options include: not at all; a little; quite a bit; very much.
change in quality of life measured via the ECHO EXERT survey | 3 Months
  The Experience of Care and Health Outcomes (ECHO) Survey asks three questions about participant experience with the exercise intervention. Response options include: not at all; not much; mixed; somewhat; very much so.
change in quality of life measured via the Health Belief Scale | 3 Months
  The Health Belief Scale asks questions regarding exercise therapy. Response options include: strongly disagree - strongly agree, where 1 equals strongly disagree and 4 equals strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Sturgeon, PhD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/56/NCT03905356/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT03905356/ICF_001.pdf